CLINICAL TRIAL: NCT00471432
Title: A Phase I Study of a Second Generation Clusterin Antisense Oligonucleotide (OGX-011) in Combination With Docetaxel
Brief Title: OGX-011 and Docetaxel in Treating Patients With Metastatic or Locally Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I154; CAN-NCIC-IND154 (Other: PDQ); ONCOGENEX-OGX-01-02 (Other: Oncogenex Technologies); CDR0000547039 (Other: PDQ)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer; Breast Cancer; Kidney Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent prostate cancer; stage IV prostate cancer; recurrent renal cell cancer; stage IV renal cell cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent bladder cancer; stage IV bladder cancer; recurrent breast cancer; stage IV breast cancer; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; unspecified adult solid tumor, protocol specific; male breast cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Kidney Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: custirsen sodium
Drug: docetaxel
Other: pharmacological study

SUMMARY:
RATIONALE: OGX-011 may kill tumor cells by blocking some of the proteins that may cause tumor cells to grow. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving OGX-011 together with docetaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of OGX-011 when given together with docetaxel in treating patients with metastatic or locally recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and recommended phase II dose of OGX-011 when administered with docetaxel in patients with metastatic or locally recurrent solid tumors.

Secondary

* Determine the pharmacokinetic profile of this regimen in these patients.
* Assess the effect of OGX-011 on serum clusterin levels and clusterin expression in peripheral blood mononuclear cells and accessible tumors.
* Assess objective response in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter, dose-escalation study of OGX-011. Patients are sequentially assigned to 1 of 2 treatment schedules.

* Schedule A: Patients receive OGX-011 IV over 2 hours on days 1, 3, 5, 8, 15, 22, 29, and 36 of course 1 and once weekly in weeks 1-6 of all subsequent courses. Patients also receive docetaxel IV over 1 hour once weekly in weeks 1-5. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Schedule B: Patients receive OGX-011 IV over 2 hours on days -7, -5, -3, 1, 8, and 15 of course 1 and days 1, 8, and 15 of all subsequent courses. Patients also receive docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks (course 1 is 4 weeks in duration) for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of OGX-011 (in each schedule) until the recommended phase II dose (RPTD) is determined. The RPTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients undergo serum collection periodically for pharmacokinetic and pharmacodynamic analysis.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumors that have been shown to overexpress clusterin, including but not limited to, any of the following:

  * Prostate cancer
  * Renal cell carcinoma
  * Non-small cell lung cancer
  * Bladder cancer
  * Breast cancer
  * Ovarian cancer
* Metastatic or locally recurrent disease
* Refractory to standard curative therapy or no standard curative therapy exists

  * Patients with prostate cancer must be hormone refractory (i.e., have documented evidence of progression while receiving androgen ablative therapy)
* Measurable or nonmeasurable disease

  * Measurable disease defined as measurable lesion ≥ 20 mm by x-ray, physical exam, or nonspiral CT scan or ≥ 10 mm by spiral CT scan
* No documented CNS metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* Creatinine ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* PT/INR and PTT normal
* No uncontrolled pain
* No known bleeding disorder
* No history of serious allergic reaction to taxane (paclitaxel or docetaxel)
* No preexisting peripheral neuropathy ≥ grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious illness or medical conditions that would preclude study compliance, including any of the following:

  * Active uncontrolled infection
  * Significant cardiac dysfunction
* No significant neurological disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* No prior strontium chloride Sr 89
* No more than 2 prior chemotherapy regimens, including adjuvant or neoadjuvant chemotherapy (for patients assigned to schedule B [docetaxel once every 3 weeks])
* More than 4 weeks since prior chemotherapy and recovered
* At least 4 weeks since prior antiandrogens
* More than 4 weeks since prior external-beam radiotherapy, except low-dose nonmyelosuppressive radiotherapy
* No prior radiotherapy to ≥ 30% of marrow-bearing areas (for patients assigned to schedule B [docetaxel once every 3 weeks])
* At least 28 days since prior new anticancer therapy
* At least 28 days since prior and no other concurrent investigational agents
* No concurrent radiotherapy, except low-dose nonmyelosuppressive radiotherapy
* No other concurrent cytotoxic therapy
* Concurrent luteinizing hormone-releasing hormone agonist allowed (if already initiated in patients with prostate cancer)
* No concurrent anticoagulant therapy (i.e., heparin, warfarin)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-04-04 (Actual); Primary Completion 2006-03-09 (Actual); Study Completion 2009-12-21 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity
Recommended phase II dose of OGX-011

SECONDARY OUTCOMES:
Pharmacokinetic profile
Serum clusterin levels and clusterin expression in peripheral blood mononuclear cells and accessible tumors
Objective response

CONTACTS AND LOCATIONS:
Overall Officials: Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chi KN, Siu LL, Hirte H, Hotte SJ, Knox J, Kollmansberger C, Gleave M, Guns E, Powers J, Walsh W, Tu D, Eisenhauer E. A phase I study of OGX-011, a 2'-methoxyethyl phosphorothioate antisense to clusterin, in combination with docetaxel in patients with advanced cancer. Clin Cancer Res. 2008 Feb 1;14(3):833-9. doi: 10.1158/1078-0432.CCR-07-1310. PMID 18245546